CLINICAL TRIAL: NCT00369473
Title: A Long-Term Assessment of Safety and Physical Function With AMG 108 Subcutaneous Monthly Treatment in Subjects With Rheumatoid Arthritis
Brief Title: Long-Term Assessment of Safety and Physical Function With AMG 108 in RA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20060119
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — AMG 108

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): 350
  Interventions: Drug: AMG 108
- 2 (Experimental): 350
  Interventions: Drug: AMG 108

INTERVENTIONS:
Drug: AMG 108 — 125 mg via SC (subcutaneous) injection every 4 weeks
  Arms: 1
Drug: AMG 108 — 250 mg via SC (subcutaneous) injection every 4 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to assess long-term safety of SC AMG 108 in the treatment of RA

ELIGIBILITY:
Inclusion Criteria:

* Only subjects eligible for and completing 24 weeks of study 20050168 will be permitted to enroll.

Exclusion Criteria:

* Subjects not eligible for or not completing 24 weeks of study 20050168 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To assess long-term safety of AMG 108 SC in subjects with RA previously enrolled in study 20050168 | 144 Weeks

SECONDARY OUTCOMES:
To determine whether long-term use of AMG 108 improves function in subjects with RA | 144 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com